CLINICAL TRIAL: NCT03329209
Title: An Open-Label, Single-Center, Phase 1 Study to Determine the Pharmacokinetics of Single Intravenous Dose of Vedolizumab 300 mg in Healthy Adult Chinese Subjects
Brief Title: A Study to Determine the Pharmacokinetics (PK) of Single Intravenous (IV) Dose of Vedolizumab 300 Milligram (mg) in Healthy Adult Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Vedolizumab-1014; U1111-1197-3577 (Registry Identifier: WHO)
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Colitis, Ulcerative; Crohn Disease
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, infusion, intravenously over 30-minutes, once on Day 1.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion.

SUMMARY:
The purpose of this study is to assess the PK of vedolizumab following a single intravenous infusion in healthy adult Chinese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab is being tested to treat people who have ulcerative colitis (UC) or Crohn's disease (CD). This study will look at the PK, safety, and tolerability of vedolizumab following a single intravenous infusion of vedolizumab IV in healthy adult Chinese participants.

The study will enroll approximately 16 participants. All participants will be assigned to receive a single dose of vedolizumab IV 300 mg on Day 1.

This single center trial will be conducted in China. The overall time to participate in this study is approximately 7 months. Participants will make multiple visits to the clinic, and will be contacted by telephone, 6 months after single dose of study drug for a follow-up safety survey assessment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 19.0 to 26.0 kilogram per square meter (kg/m^2) inclusive at Screening.

Exclusion Criteria:

1. Has one or more positive response on the progressive multifocal leukoencephalopathy (PML) subjective symptoms checklist at Screening or before dosing on Day 1.
2. Has had a surgical procedure requiring general anesthesia within 30 days before the initial Screening Visit or is planning to undergo a surgery that requires general anesthesia during the study period (through Final Visit/Day 127).
3. For participants who are negative for hepatitis B surface antigen (HBsAg) but are positive for either surface antibodies and/or core antibodies, hepatitis B virus Deoxyribonucleic Acid (DNA) polymerase chain reaction will be performed and any result that meets or exceeds detection sensitivity will be excluded.
4. Has poor peripheral venous access.
5. Has a QT interval with Fridericia correction method (QTcF) greater than (>) 430 millisecond (ms) (males) or >450 ms (females) or PR outside the range 120 to 220 ms, confirmed with 1 repeat testing within a maximum of 5 minutes, at the Screening Visit or Check-in (Day -1).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in China from 05 March 2018 to 05 September 2018.
Pre-assignment Details: Healthy Chinese participants were enrolled to receive a single dose of vedolizumab intravenous 300 milligram (mg).
Period: Overall Study
Arm/Group | Vedolizumab 300 mg
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled and received 1 dose of study drug.
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 16
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 167.00 (7.474)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 63.83 (6.448)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 22.87 (1.622)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Serum Concentration for Vedolizumab
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: The pharmacokinetic (PK) analysis set consisted of all participants who received study drug and had at least 1 measurable serum concentration.
Measure: Geometric Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 16
microgram per milliliter (mcg/mL) | 136.4120 (15.90597)

2. Primary Outcome: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Vedolizumab
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: The PK analysis set consisted of all participants who received study drug and had at least 1 measurable serum concentration.
Measure: Geometric Mean (Standard Deviation); unit: day*microgram per milliliter(day*mcg/mL)
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 16
day*microgram per milliliter(day*mcg/mL) | 2342.5803 (294.75822)

3. Primary Outcome: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Vedolizumab
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 16
day*mcg/mL | 2377.6463 (296.46345)

4. Secondary Outcome: Percentage of Participants With Positive Anti-vedolizumab Antibody (AVA)
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: The safety analysis set consisted of all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 16
percentage of participants | 37.5

5. Secondary Outcome: Percentage of Participants With Positive Neutralizing AVA
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: The safety analysis set consisted of all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Vedolizumab 300 mg
Number analyzed (Participants) | 16
percentage of participants | 37.5

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAE) are adverse events that started after the infusion of study drug and no more than Day 127
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report AES occurring at any other time during the study. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab 300 mg (N=16)
Upper respiratory tract infection (Infections and infestations) | 4
Blood creatine phosphokinase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Leukocyturia (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03329209/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03329209/SAP_001.pdf